CLINICAL TRIAL: NCT04691531
Title: Decreasing the Invasiveness of Ultrasound Guided Caudal Block: A Randomized Controlled Trial Comparing Between 22-gauge and 27-guage Needles
Brief Title: Decreasing the Invasiveness of Ultrasound Guided Caudal Block: A Comparison Between 22-gauge and 27-guage Needles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, omar ahmad ababneh, Principal investigator, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4599/2020/67
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Anesthesia; Pain; Caudal Block; Pediatric Anesthesia; Abdominal Surgeries
Keywords: Caudal block; Ultrasound; Pediatric anesthesia; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group C (Experimental): After induction of general anesthesia, patients will undergo caudal block by classical Gauge 22 needle under ultrasound guidance using a linear probe 5.5-12 MHz, and Bupivacaine 1 ml/kg of 0.25% will be injected.
  Interventions: Device: The use of classical Gauge 22 needle
- Group S (Experimental): After induction of general anesthesia, patients will undergo caudal block by Gauge 27 needle under ultrasound guidance using a linear probe 5.5-12 MHz, and Bupivacaine 1 ml/kg of 0.25% will be injected.
  Interventions: Device: The use of classical Gauge 27 needle

INTERVENTIONS:
Device: The use of classical Gauge 22 needle — After induction of general anesthesia, patients will undergo caudal block by using classical Gauge 22 needle under ultrasound guidance using a linear probe 5.5-12 MHz.
  Arms: group C
Device: The use of classical Gauge 27 needle — After induction of general anesthesia, patients will undergo caudal block by using Gauge 27 needle under ultrasound guidance using a linear probe 5.5-12 MHz.
  Arms: Group S

SUMMARY:
Ultrasound (US) has facilitated the use of caudal block in children and visualization of the needle during insertion. This prospective clinical trial study compares between two different sizes of the used needles, in terms of success rate, number of punctures, detection of the US signs (visualization of the needle, dural displacement, turbulence, and distention), and complications in pediatrics aging between 6-36 months requiring elective lower abdominal and perineal surgeries.

DETAILED DESCRIPTION:
Ultrasound (US) has facilitated the use of caudal block in children, allowing an initial assessment of the anatomy of the sacrum, including the relationship of the sacral hiatus to the dural sac ending. Real-time US allows visualization of the needle during insertion to reach the dural sac, and to see the turbulence and distention of the layers during injection of the local anesthetic drug.

This prospective clinical trial study compares between two different sizes of the used needles, in terms of success rate, number of punctures, detection of the US signs (visualization of the needle, dural displacement, turbulence, and distention), and complications in pediatrics aging between 6-36 months requiring elective lower abdominal and perineal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 months and 36 months
* Undergoing elective lower abdominal or perineal surgeries

Exclusion Criteria:

* Refusal of the legal guardian of the patient.
* Patients aging less than 6 months, or older than 36 months.
* Emergency surgeries.
* Coagulopathy.
* infection at the site of procedure.
* Uncorrected hypovolemia.
* Increased intracranial pressure.
* Congenital anomalies at the site of procedure.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Opioids requirements intraoperatively | 90 minutes
  The investigators will document the required dose of opioids intraoperatively
Pain score in the post-anesthesia care unit (PACU) | 120 minutes
  Pain score will be assessed regularly during the stay in the PACU using a pain scoring scale, where the score is interpreted from 0 to 10, in which 0 means no pain and 10 signifies very severe pain.
Peri-operative complications | 210 minutes
  Peri-operative complications related to the caudal block procedure will be documented from the start of the procedure till the discharge from the post-anesthesia care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jordan